CLINICAL TRIAL: NCT04861883
Title: A Diagnostic Test Study of Characteristic Sound Waves in the Middle and Third Trimester of Pregnancy Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, dean of orthopedic department, Qianfoshan Hospital
Other Study IDs: SFUYIN-05
Record Dates: First submitted 2021-03-14; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Pregnancy; Radial Artery
Keywords: pregnancy; diagnostic test; sound waves; radial artery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 76 healthy the Middle and Third Trimester pregnant women in the trial group: The pulse sound waves of three parts and five layers of each of the two hands of 76 pregnant women will be collected by Pulse Detection System of Sound Waves.
- 76 relatively healthy non-pregnant women in the control group: The pulse sound waves of three parts and five layers of each of the two hands of 76 relatively healthy non-pregnant women will be collected by Pulse Detection System of Sound Waves.

SUMMARY:
Pregnancy is a very complex and coordinated physiological process.The physiological changes are closely related to the physiological function of Zang-fu organs, which leads to the change of slippery pulse. By touching different levels of depth and the part of the radial artery, it is found that the formation mechanism of pulse information, especially unsmooth pulse, is similar to the principle of sonar emission and reception: the heart is equivalent to the transmitting device of sonar wave. Each contraction of the heart produces a cluster of powerful sound waves, which are rapidly transmitted to the whole body along the arterial wall and the blood in it as a medium. More than 90% of the arterial blood flow of normal organs and tissues is a steady laminar flow, which does not produce turbulence, so there is abnormal vibration when a certain organ and tissue has pathological changes. The arterial blood flow is squeezed and deformed which causing turbulence and abnormal vibrations, which are fused with a larger cluster of sound waves transmitted by the heart and then transmitted to the whole body. The investigators can feel this kind of sound waves which combine abnormal vibration waves by touching different levels of arteries close to the body surface, including the radial artery. At the same time, Professor Lucheng Song's team has conducted in-depth research on the characteristic unsmooth pulse of stable coronary heart disease, liver cirrhosis, gastritis and other diseases.During pregnancy, due to the significant increase in blood flow and maternal changes , the shape of sound waves transmitted to the radial artery in the artery will be changed. Professor Lucheng Song found in clinical practice that the pregnant pulse will have different sensations of smoothness and penetration in different parts of the finger, by touching different levels of depth and the part of the radial artery. It was found that the pulse condition of normal pregnant women in the middle and third trimester of pregnancy was different from that of normal non-pregnant women in different level and part of radial artery.This study will verify the efficacy of pulse diagnosis of traditional Chinese medicine in the diagnosis of pregnancy and lay a foundation for the diagnosis of abnormal pregnancy.

DETAILED DESCRIPTION:
Pregnancy is a special physiological stage for women, and the changes of Qi and blood in the body can be reflected in time by the dynamic changes of pulse, which provides an important basis for clinical diagnosis and treatment. Pregnancy is a very complex and coordinated physiological process, in which the physiological changes related to pulse changes include: 1. Changes in blood pressure. Relatively speaking, in the middle trimester, the blood pressure is low; at the end of the pregnancy, the blood pressure increases slightly, the general systolic blood pressure does not change, the diastolic blood pressure decreases slightly due to peripheral vasodilation, hemodilution and placental arteriovenous short circuit, and the pulse pressure increases slightly. 2.The change of cardiac output. Cardiac output increases gradually from 8-10 weeks of gestation and reaches the peak at 32-34 weeks of pregnancy until delivery. 3.The change of blood volume. The maternal blood volume begins to increase from 6-8 weeks of pregnancy and reaches the peak at 32-34 weeks of pregnancy until delivery. The above physiological changes are closely related to the physiological function of Zang-fu organs, which leads to the change of slippery pulse. With the continuous development of modern pulsology, Professor Lucheng Song has been studying the knowledge of modern physics such as hemodynamics, hydrodynamics and acoustics based on his long-term clinical practice. By touching different levels of depth and the part of radial artery, it is found that the formation mechanism of pulse information, especially unsmooth pulse, is similar to the principle of sonar emission and reception: the heart is equivalent to the transmitting device of sonar wave. Each contraction of the heart produces a cluster of powerful sound waves, which are rapidly transmitted to the whole body along the arterial wall and the blood in it as a medium.More than 90% of the arterial blood flow of normal organs and tissues is a steady laminar flow, which does not produce turbulence, so there is abnormal vibration when a certain organ and tissue has pathological changes. The arterial blood flow is squeezed and deformed which causing turbulence and produces abnormal vibrations, which are fused with a larger cluster of sound waves transmitted by the heart and then transmitted to the whole body. The investigators can feel this kind of sound waves which combine abnormal vibration waves by touching different levels of arteries close to the body surface, including the radial artery. At the same time, Professor Lucheng Song's team has conducted in-depth research on the characteristic unsmooth pulse of stable coronary heart disease, liver cirrhosis, gastritis and other diseases.Different pulse sound waves were collected by using Pulse Detection System of Sound Waves(PDSSW),and ideal results were obtained through analysis. During pregnancy, due to the significant increase in blood flow and maternal changes,the shape of sound waves transmitted to the radial artery in the artery will be changed. Professor Lucheng Song found in clinical practice that the pregnant pulse will have different sensations of smoothness and penetration in different parts of the finger, by touching different levels of depth and the part of the radial artery. It was found that the pulse condition of normal pregnant women in the middle and third trimester of pregnancy was different from that of normal non-pregnant women in different level and part of radial artery.Based on the above analysis, this study will use PDSSW to collect the pulse waves of 76 the Middle and Third Trimester of Pregnancy and 76 relatively healthy women.Fourier transform, wavelet analysis, Hilbert-Huang transform and other methods will be used to identify the different characteristics of the sound wave signals, and observe the time-frequency domain characteristics of the trial group and the control group. Then diagnostic tests will be performed to calculate the sensitivity and specificity of PDSSW in the diagnosis of the middle and third trimester of pregnancy women.This trial will further verify the effectiveness of pulse diagnosis and lay a foundation for the diagnosis of complication of pregnancy by pulse diagnosis instruments.

ELIGIBILITY:
Inclusion Criteria:

Trial group:

1. The pregnant women in the middle and third trimester of pregnancy diagnosed by laboratory and B-ultrasound；
2. The first singleton pregnancy, from 13 weeks to parturition；
3. There are no pregnancy complications, the vital signs are stable, and the biochemical examination is normal;
4. Patients who have informed consent to accept this pulse collection.

Control group:

1. Those who are included in the relatively healthy population are those with negative diagnostic criteria for early pregnant women;
2. Patients who have informed consent to accept this pulse collection;
3. The vital signs are stable, the biochemical tests are normal, and there are no severe brain, liver and kidney diseases.

Exclusion Criteria:

Trial group:

1. Pregnant women with ovarian, fallopian tube, uterine diseases, hypertension and diabetes during pregnancy;
2. Definitely diagnosed patients with respiratory, cardiovascular, cerebrovascular, liver and kidney, blood, endocrine and other system diseases and severe infectious diseases;
3. Those who have had a cesarean section or history of miscarriage;
4. Those who have a serious illness and sit for less than 10 minutes in a quiet state;
5. Patients with mental illness, depression, and cognitive impairment;
6. Those who are not easy to collect pulse manifestation such as pulse on back of wrist and oblique-running pulse;
7. Those who have incomplete information due to subjective or objective reasons that affect the result judgment;
8. Patients with Parkinson's or other limb tremors.

Control group:

1. Those who have had a history of miscarriage or ectopic pregnancy;
2. Patients with severe infectious diseases;
3. Those who are not easy to collect pulse manifestation such as pulse on back of wrist and oblique-running pulse;
4. The incomplete information affects the judgment of the result due to subjective or objective reasons;
5. Patients with Parkinson's or other limb tremors;
6. Menstrual women.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The middle and third trimester Pregnant women and relatively healthy non-pregnant women
Sampling Method: Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-03-09 (Estimated); Study Completion 2022-03-09 (Estimated)

PRIMARY OUTCOMES:
Frequencies of characteristic sound waves in the pulses | The data will be collected,analyzed and calculated in about 7 days.
  Using the Pulse Detection System of Sound Waves (PDSSW) to collect the pulse waves of both hands. The percentage(%) of frequencies of characteristic sound waves in the pulse will be calculated.
The changes of sound waves in the pulses | The discovery of characteristic sound waves may take 3 months.
  The changes of sound waves in the middle and third trimester of pregnancy women at different hertz(Hz) frequencies and SMPL amplitudes will be compared with relatively healthy women's.
Diagnostic test | Diagnostic tests may take about 1 month.
  The Percentage(%) of specificity, sensitivity, positive likelihood ratio and negative likelihood ratio of the "Pulse Detection System of Sound Waves" in the diagnosis of the middle and third trimester of pregnancy women.
Sound waves analysis | 1 month
  The Hertz(Hz) of the different segments of the sound waves in Wavelet transform; The Hertz(Hz) of the different layers of the sound waves in Hilbert-Huang; The SMPL amplitudes of sound waves in Discrete Fourier Transform； The sample Entropy(sampEn) of sound waves in Sample Entropy.

CONTACTS AND LOCATIONS:
Overall Officials: Lucheng Song, Doctor, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

REFERENCES:
- [Background] Cui H, Su J, Liang WW, Wang HL, Wang HF. Diagnostic analysis of abnormal increase of PASP in fetus in middle- and late-stage pregnancy by color Doppler echocardiography. Br J Radiol. 2020 Jun;93(1110):20191011. doi: 10.1259/bjr.20191011. Epub 2020 Mar 25. PMID 32160003
- [Background] Rodriguez C, Chi YY, Chiu KH, Zhai X, Lingis M, Williams RS, Rhoton-Vlasak A, Nichols WW, Petersen JW, Segal MS, Conrad KP, Mohandas R. Wave reflections and global arterial compliance during normal human pregnancy. Physiol Rep. 2018 Dec;6(24):e13947. doi: 10.14814/phy2.13947. PMID 30578623
- [Background] Li K, Zhang S, Chi Z, Yang Y, Jiang H, Yang L, Wang A, Zhang L, Chen F, Zheng D. Arterial Pulse Waveform Characteristics Difference between the Three Trimesters of Healthy Pregnant Women. Annu Int Conf IEEE Eng Med Biol Soc. 2018 Jul;2018:5317-5320. doi: 10.1109/EMBC.2018.8513492. PMID 30441537
- [Background] Li K, Zhang S, Yang L, Jiang H, Chi Z, Wang A, Yang Y, Li X, Hao D, Zhang L, Zheng D. Changes of Arterial Pulse Waveform Characteristics with Gestational Age during Normal Pregnancy. Sci Rep. 2018 Oct 22;8(1):15571. doi: 10.1038/s41598-018-33890-1. PMID 30349022
- [Background] Martin JN Jr, Tucker JM. Missing or making the timely diagnosis of acute fatty liver of pregnancy (AFLP): lessons learned. J Matern Fetal Neonatal Med. 2022 Sep;35(18):3595-3601. doi: 10.1080/14767058.2020.1832075. Epub 2020 Oct 9. PMID 33032483
- [Background] Rodger M, Sheppard D, Gandara E, Tinmouth A. Haematological problems in obstetrics. Best Pract Res Clin Obstet Gynaecol. 2015 Jul;29(5):671-84. doi: 10.1016/j.bpobgyn.2015.02.004. Epub 2015 Mar 4. PMID 25819750
- [Background] Lumbers ER, Pringle KG. Roles of the circulating renin-angiotensin-aldosterone system in human pregnancy. Am J Physiol Regul Integr Comp Physiol. 2014 Jan 15;306(2):R91-101. doi: 10.1152/ajpregu.00034.2013. Epub 2013 Oct 2. PMID 24089380
- [Background] Bilton K, Hammer L, Zaslawski C. Contemporary Chinese pulse diagnosis: a modern interpretation of an ancient and traditional method. J Acupunct Meridian Stud. 2013 Oct;6(5):227-33. doi: 10.1016/j.jams.2013.04.002. Epub 2013 Apr 24. PMID 24139459
- [Background] Drukker L, Droste R, Chatelain P, Noble JA, Papageorghiou AT. Safety Indices of Ultrasound: Adherence to Recommendations and Awareness During Routine Obstetric Ultrasound Scanning. Ultraschall Med. 2020 Apr;41(2):138-145. doi: 10.1055/a-1074-0722. Epub 2020 Feb 27. PMID 32107757